CLINICAL TRIAL: NCT04156126
Title: Measuring Markers of Immune Tolerance to Predict Women at Risk of Miscarriage or Failed Embryo Transfer Prior to Symptoms
Brief Title: Measuring Immune Tolerance to Predict Miscarriage or Failed Embryo Transfer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Chandra C. Shenoy, Assistant Professor of Obstetrics and Gynecology, Mayo Clinic
Other Study IDs: 18-011413
Record Dates: First submitted 2019-08-12; First posted 2019-11-07 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Infertility; Pregnancy Loss; Spontaneous Abortion
MeSH Terms: conditions — Infertility; Abortion, Spontaneous | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In cohort 1, 10mL blood samples will be drawn from subjects undergoing a frozen embryo transfer at 4 different time points.
  In cohort 2, 10mL blood samples will be drawn from subjects with spontaneous conception at 1 time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infertility - Frozen Embryo Transfer: Adult females undergoing a frozen embryo transfer
  Interventions: Other: Blood Collection
- Spontaneous Conception: Adult females presenting with positive pregnancy test to the Obstetrics Department
  Interventions: Other: Blood Collection

INTERVENTIONS:
Other: Blood Collection — Blood Collection

SUMMARY:
Pregnancy is a unique period which requires alterations in the immune system to allow for tolerance of a haploidentical fetus. The goal of this study is to measure maternal blood levels of proteins known to promote immune tolerance in early implantation and pregnancy to look for associations between tolerance, miscarriage and failed embryo transfer. Establishing predictive factors of miscarriage and failed in vitro fertilization could have implications for a large portion of couples and serve to guide current and future family planning efforts.

DETAILED DESCRIPTION:
There is increasing evidence of the importance of T cell immunoglobulin and mucin-containing protein 3 (Tim-3) in suppressing allograft rejection, and thus it is hypothesized to play a role in pregnancy. Galectin-9 (Gal-9) is a ligand for Tim-3 activation which promotes Th1 apoptosis signaling. Activation of Tim-3 by Gal-9 has also been shown to suppress NK cell cytotoxicity at the maternal-fetal interface. Previous studies have evaluated Tim-3 expression on NK cells in the first trimester and found in comparison to normal pregnancies, patients with recurrent miscarriage had decreased Tim-3 expression and less anti-inflammatory cytokine production. In a mouse model, transfer of Tim-3 expressing NK cells reduced miscarriage rates. During the first trimester, Gal-9 levels increase and remain elevated throughout pregnancy. Preliminary data in a small population of patients who had miscarriages were found to have significantly lower Gal-9 levels detected at 8 weeks gestation compared to those who continued on to have a term pregnancy. Additionally there is evidence that Gal-9 increases production of interleukin (IL-4), and in patients with recurrent miscarriage IL-4 levels are decreased [5]. These identifications have prompted further investigation into predictive value of Gal-9 and IL-4 levels in early pregnancy on the outcome of a pregnancy.

Angiogenic factors, such as vascular endothelial growth factors (VEGF), have been shown to have a critical role in pregnancy at both the local and systemic level. Locally, CD56+ uterine natural killer cells within the endometrium express higher levels of VEGF in women with recurrent miscarriage versus women with proven fertility. Histological differences in VEGF expression and placental vascular bed patterns have been observed in tissue from patients with a miscarriage compared to women with a viable pregnancy. Serum VEGF levels are significantly different in patients with recurrent pregnancy loss than in women with proven fertility [8]. Serum VEGF levels, including VEGF-A, -C, and -D, are significantly higher at 8 weeks gestation in pregnancies that result in a spontaneous loss compared to pregnancies that go on to result in a live birth. Therefore, additional studies are needed to establish if early first trimester serum levels of VEGFs, Gal-9, and IL-4 are significantly different in pregnancies that result in miscarriage or live birth. Miscarriage affects approximately 15-20% of pregnancies. Therefore, establishing predictive factors of miscarriage could have implications for a large portion of couples and could serve to guide current and future family planning efforts. It is, essential to gain an understanding of mechanisms underlying infertility and miscarriage, so that more effective treatments and protocols can be developed.

The study hypothesis states low levels of Gal-9 and IL-4, and high levels of VEGF at the time of embryo transfer will be predictive of failed embryo transfer and spontaneous miscarriage. The primary endpoint is the maternal blood levels of galectin-9, IL-4 and VEGF-A,-C,-D on the day of embryo transfer in cycles that result in live birth versus no live birth, or that result in miscarriage compared to live birth.

ELIGIBILITY:
Inclusion Criteria:

* Females, 18 years old or older
* Patients undergoing a frozen embryo transfer OR confirmed intrauterine pregnancy between 5 0/7 weeks and 9 6/7 weeks gestation
* Patients planning to have all bloodwork done at Mayo Clinic Rochester
* Patients planning to deliver at Mayo Clinic or within the Mayo Clinic Health Systems

Exclusion Criteria:

* Non English speaking
* Pregnancy with multiple fetuses
* Patient has non-viable pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females age 18 or older
Study Population: Females age 18 or older who are undergoing a frozen embryo transfer or have a confirmed intrauterine pregnancy between 5 0/7 weeks and 9 6/7 week gestation.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Spontaneous Conception Cohort: change in immune tolerance, as measured by Enzyme Linked Immunosorbent Assay (ELISA) | Baseline (6-12 weeks gestation)
  Tolerance markers galectin-9, IL-4 and VEGF (-A,-B,-C,-D) will be measured for their concentration in maternal blood in women who conceived naturally, as determined by experimental standard curves.
Infertility Cohort: change in immune tolerance, as measured by Enzyme Linked Immunosorbent Assay (ELISA) | Change from baseline (day of transfer) at Day 11
  Tolerance markers galectin-9, IL-4 and VEGF (-A,-B,-C,-D) will be measured for their concentration in maternal blood in women who undergo embryo transfer, as determined by experimental standard curves.

CONTACTS AND LOCATIONS:
Overall Officials: Chandra C Shenoy, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States